CLINICAL TRIAL: NCT02852408
Title: Unintentional Liver Cauterization Increases the Postoperative Pain After Laparoscopic Cholecystectomy: A Prospective Controlled Blinded Trial
Brief Title: Liver Cauterization Increases the Postoperative Pain After Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih Basak, Dr., Umraniye Education and Research Hospital
Other Study IDs: LAP-COL-CAUTER
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Study: liver cauterized during laparoscopic cholecystectomy.
  Interventions: Procedure: Laparoscopic cholecystectomy
- Control: liver not-cauterized during laparoscopic cholecystectomy.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy

SUMMARY:
Laparoscopic cholecystectomy is a common accepted surgical operation with lower morbidity all over the world for gallstone. Although it has low morbidity, postoperative pain is challenging situation like every other operation.

DETAILED DESCRIPTION:
Postoperative pain after laparoscopic cholecystectomy has a three component: parietal, visceral and referring (shoulder) pain. Although intensities of them can be various, all of them affects the total pain together. Unintentional liver cauterization during laparoscopic cholecystectomy is unwanted, but sometimes unavoidable complication/process. However its effect on postoperative pain is not studied with detail in literature.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II
* Presumptive diagnosis of benign gallbladder disease

Exclusion Criteria:

* The patients with concurrent chronic disease like osteoporosis, and liver, pulmonary or renal disease, malignant disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have scheduled for laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) abdominal pain scores | Postoperative 2nd hour
Visual analog scale (VAS) abdominal pain scores | Postoperative 24th hour